CLINICAL TRIAL: NCT04420455
Title: The Effects of Enoximone in Acute Exacerbation COPD
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: A limited number of inclusions due to the Covid-pandemic
Sponsor: Rijnstate Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-1432
Record Dates: First submitted 2020-01-31; First posted 2020-06-09 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2021-12

CONDITIONS: COPD Exacerbation; Enoximone; Phosphodiesterase Inhibitor
MeSH Terms: interventions — Enoximone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Enoximone (Experimental): Patients will receive three times a dose of 0.5 mg/kg enoximone with a one-hour-interval.
  Interventions: Drug: Enoximone

INTERVENTIONS:
Drug: Enoximone — Patients will receive three times a dose of 0.5 mg/kg enoximone with a one-hour-interval.

SUMMARY:
Introduction:

The pharmacodynamic properties of enoximone could be beneficial for patients with an Acute Exacerbation COPD (AE-COPD). This research will focus on patients suffering of a severe AE-COPD and the bronchodilatory and inotropic effects of lower doses of enoximone. The main objective of the pilot study is to investigate if there is a bronchodilatory effect of enoximone in patients with AE-COPD. Secondary objective is to investigate a dose responsiveness in a range between 0.5 and 1.5 mg/kg enoximone.

Methods:

The study design is a prospective interventional non-randomized clinical series study involving patients admitted and intubated at the Intensive Care Unit (ICU) with an AE-COPD. Patients will receive three times a dose of 0.5 mg/kg enoximone with a one-hour-interval. The primary objective is a reduction in auto-positive end-expiratory pressure (PEEP) after enoximone compared to baseline. A dose-titration will test for dose dependency. Secondary objectives are a reduction in ventilator pressures, a reduction in pulmonary artery pressures and an increase in cardiac output.

DETAILED DESCRIPTION:
Ventilator will be set during the study period at Volume Controle, 6 ml/kg, 5 PEEP and a respiratory rate of 15 bpm with an I:E-ratio of 1:2.

Salbutamol/ipratropium bromide and magnesium sulphate will be administered at baseline (t=0h) and measurements will be made for an hour.

At T=1h the first dose of 0.5 mg/kg enoximone will be administered and will be repeated at T=2h and T=3h. Ventilator derived variables will be obtained every fifteen minutes and echocardiography, arterial and central venous bloodgas analyses every hour until t=6h.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an AE-COPD for which intubation occurred within 24 hours before enrolment.

Exclusion Criteria:

* Patients with known asthma or interstitial lung disease (ILD)
* Known neurodegenerative diseases such as Amyotrophic Lateral Sclerosis (ALS), Multiple Sclerosis (MS), Guillain-Barre and Dementia
* Hypertrophic obstructive cardiomyopathy (HOCM)
* Severe aortic stenosis with aortic valve area < 1cm2
* Known ventricular arrhythmias
* Severe kidney disorders with Glomerular Filtration Rate (GFR) < 30
* Severe liver insufficiency with spontaneous PT/INR > 1.5
* Pregnancy
* Lactation
* High dose-diuretics use (daily dose of >480 mg furosemide)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2020-05-12 (Actual); Primary Completion 2021-12-21 (Actual); Study Completion 2021-12-21 (Actual)

PRIMARY OUTCOMES:
PEEP | within 6 hoursmeasured every 15 minutes
  Reduction in intrinsic PEEP, in cmH2O

SECONDARY OUTCOMES:
Lung compliance | within 6 hours, measured every hour
  ml/H2O
Airway resistence | within 6 hours, measured every hour
  cmH2O/L/sec
VEI | within 6 hours, measured every hour
  ml
VCO2 | within 6 hours, measured every hour
  ml/min
etCO2 | within 6 hours, measured every hour
  kPa
Vd/Vt | within 6 hours, measured every hour
  Measured by Bohr-equation, in percentage
FiO2 | within 6 hours, measured every hour
  percentage
Shunt fraction | within 6 hours, measured every hour
  measured by Fick-equation, using the SvO2, in percentage
Cardiac Output | within 6 hours, measured every hour
  Measured by echocardiography (LVOT VTI), ml/hr
RVSP | within 6 hours, measured every hour
  Measured by echocardiography, in mmHg
TAPSE | within 6 hours, measured every hour
  Measured by echocardiography, in mm
MAPSE | within 6 hours, measured every hour
  Measured by echocardiography, in mm
LV Ejection Fraction | within 6 hours, measured every hour
  Measured by echocardiography, in percentage
Bloodgas analysis | within 6 hours, measured every hour
  Arterial bloodgas analysis and central venous gas analysis (through catheter placed in superior vena cava)

CONTACTS AND LOCATIONS:
Locations (1):
- M.V. Koning, Arnhem, M, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF, CSR
Time Frame: after publication
Access Criteria: upon reasonable request, available by the researchers